CLINICAL TRIAL: NCT07126886
Title: A Multicenter, Prospective, Clinical Trial Evaluating a Single Layer Amniotic Membrane and Standard of Care Versus Matched Controls in the Management of Nonhealing Pressure Ulcers
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Applied Biologics, LLC (Industry)
Collaborators: SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XPURT
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pressure Ulcer; Ulcer, Pressure; Pressure Wound; Pressure Area
MeSH Terms: conditions — Pressure Ulcer | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: It is a prospective multicenter controlled clinical trial using matched controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Debridement, off-loading, reduction of bacterial burden, and proper moisture balance using dressings.
  Interventions: Other: Standard of Care
- XPURT + SOC (Experimental): Single-layer amniotic membrane plus standard of care.
  Interventions: Other: XPURT + SOC

INTERVENTIONS:
Other: Standard of Care — Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 20 weeks, whichever occurs first.
  Arms: Standard of Care
Other: XPURT + SOC — Participants will receive weekly applications of XPURT and Standard of Care until ulcer closure, or a maximum of 20 weeks, whichever occurs first.
  Arms: XPURT + SOC

SUMMARY:
A multicenter, prospective, clinical trial evaluating a single-layer amniotic membrane (XPURT) and standard of care versus matched controls in the management of nonhealing pressure ulcers.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, controlled clinical study consisting of 100 subjects from up to 30 providers. The subjects receive XPURT and SOC. The target ulcers are evaluated weekly by the investigator. The subject is treated once a week, to receive weekly applications of XPURT + SOC for up to 20 weeks or until the study ulcer has completely closed (i.e. 100% closure as assessed by the investigator and confirmed 2 weeks later at the closure confirmation visit (CCV). One additional visit per week is optional for both arms, for the purpose of changing only (1) the secondary dressing in the XPURT arm or (2) change the standard of care dressing in the control arm.

ELIGIBILITY:
Inclusion Criteria:

* The potential subject must be at least 18 years of age or older.
* The potential subject must agree to attend the weekly study visits required by the protocol.
* The potential subject must be willing and able to participate in the informed consent process.
* The potential subject must have a full thickness pressure ulcer NPIAP stage 3 through stage 4 without exposed bone of greater than or equal to one month in duration located on the trunk (sacral, trochanteric, or ischial).
* At enrollment, the potential subject must have a target ulcer with a minimum surface area of 2 cm2 and a maximum surface area of 100 cm2 measured post debridement with the imaging device.
* The potential subject has adequate off-loading of the ulcer.

Exclusion Criteria:

* The potential subject is known to have a life expectancy of < 3 months.
* The potential subject's target ulcer is not a pressure ulcer.
* The target ulcer is infected, requires systemic antibiotic therapy, or there is cellulitis in the surrounding skin.
* The target ulcer exposes tendon or bone.
* There is undermining at the wound edge or tunnelling.
* There is evidence of osteomyelitis complicating the target ulcer.
* The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing (e.g., biologics).
* The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
* The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit(For diabetics only).
* The surface area of the potential subject's target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). Imaging Device is not required for measurements taken during the historical run-in period (e.g., calculating surface area using length X width is acceptable).
* The surface area measurement of the potential subject's target ulcer decreases by 25% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (S1) to the TV-1 visit during which time the potential subject received SOC.
* The potential subject is a woman who is pregnant or considering becoming pregnant within the next 6 months.
* The potential subject has end stage renal disease requiring dialysis.
* The potential subject has participated in a clinical trial involving treatment with an investigational product within the previous 30 days.
* The potential subject, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
* The potential subject was treated with hyperbaric oxygen therapy (HBOT) or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit.
* The potential subject has a malnutrition indicator score <17 as measured on the Mini Nutritional Assessment.
* The potential subject has a known or suspected sensitivity to glutaraldehyde solutions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Complete Closure | 1-22 Weeks
  The percentage of target ulcers achieving complete wound closure in 20 weeks.

SECONDARY OUTCOMES:
Time to Healing | 1-22 Weeks
  The time to healing of the target ulcers over 20 weeks.
Percentage of Wound Area Reduction | 1-22 Weeks
  Percentage wound area reduction from TV-1 to TV-21 measured weekly with digital photographic planimetry, using an Imaging Device, and physical examination.
Adverse Events | 1-22 Weeks
  The number of product- or procedure- related adverse events.
Measure Pain | 1-22 Weeks
  Change in pain in the target ulcer assessed from TV-1 to TV-21 using the VAS scale.
Measure Quality of Life | 1-22 Weeks
  Change in quality-of-Life based on the FWS [Time Frame: TV-1, TV-4, TV-8, TV-12, TV-16, and TV-20 / Final Visit.
Measure Quality of Life | 1-22 Weeks
  Change in quality-of-Life based on the wQOL [Time Frame: TV-1, TV-4, TV-8, TV-12, TV-16, and TV-20 / Final Visit.
Average Product Usage | 1-22 Weeks
  Average number of grafts used.

CONTACTS AND LOCATIONS:
Locations (1):
- Serena Group- Monroeville, Monroeville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No